CLINICAL TRIAL: NCT03623282
Title: Study Regarding the Clinical Efficacy of Synatura® in Patients With Chronic Bronchitis Type COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ahn-Gook Pharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AG-SYN-01
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Bronchitis, COPD
Keywords: Synatura; Chronic Obstructive Pulmonary Disease; Ahn Gook Pharmaceuticals
MeSH Terms: conditions — Bronchitis; Pulmonary Disease, Chronic Obstructive | interventions — AG NPP709

STUDY DESIGN:
Intervention Model Description: Experimental(Single arm):
  The enrolled patients will be prescribed Synatura® following measurement of pre-dose pulmonary functions, quality of life and systemic inflammatory state. Pulmonary functions, quality of life and systemic inflammatory state will be repeatedly measured after taking Synatura® for 3 months, and the changes from pre-dose measurements will be observed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Synatura® 15 mL (Experimental): Synatura syrup single arm
  Interventions: Drug: Synatura® 15 mL

INTERVENTIONS:
Drug: Synatura® 15 mL — All subjects will receive Synatura® 15 mL every day three times for 3 months.
  Other Names: AG NPP709

SUMMARY:
This study aims to examine the clinical efficacy of synatura in patients with chronic bronchitis type COPD in Korea.

DETAILED DESCRIPTION:
Synatura® is a drug commonly used to suppress cough and sputum in patients with acute upper respiratory tract infection and chronic inflammatory bronchitis. According to the Phase III studies conducted in Korea, the safety and efficacy of Synatura® on antitussive and expectorant effects were confirmed in patients with acute upper respiratory infection and chronic inflammatory bronchitis. However, no studies have been conducted for the effects of Synatura® in patients with COPD. COPD is divided into emphysema type and chronic bronchitis type, while typical clinical symptoms of chronic bronchitis are cough and sputum. Therefore, Synatura®, which is effective for chronic bronchitis, is expected to be effective in patients with chronic bronchitis accompanied by COPD.

ELIGIBILITY:
Inclusion Criteria:

1. Post bronchodilator FEV1/FVC < 0.7
2. Smoking history of ≥10 packs per year
3. 40 to <75 years of age
4. Patients with symptoms of chronic bronchitis (in case they have symptoms of cough or sputum over 3 months)

Exclusion Criteria:

1. Patients with acute exacerbation
2. Patients with pneumonia
3. Patients with active tuberculosis
4. Pregnant women
5. Breast-feeding women
6. Patients with fructose intolerance

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
COPD assessment test (CAT) | Baseline, At 12weeks
  Change from Baseline in baseline to 12 weeks for COPD assessment test (CAT)

SECONDARY OUTCOMES:
Efficacy of pulmonary function in bronchitis type COPD patients | Baseline, At 12weeks
  Pulmonary function test will be performed before and 3 months after taking Synatura.
  Assessment Tools: FVC (L), FVC (%), FEV1 (L), FEV1 (%), FEV1/FVC (%), TLC (%), RV (%), RV/TLC (%), DLCO (%), DLCO/VA (%)
Efficacy of inflammation throughout the body in bronchitis type COPD patients | Baseline, At 12weeks
  Blood samples will be taken before and 3 months after taking Synatura, then stored and measured by ELISA in the laboratory.
  Assessment Tools: CRP, Fibrinogen, IL-6, TNF-α
Total number of Bronchitis Severity Score (BSS) | Baseline, At 12weeks
  Bronchitis Severity Score (BSS) will be performed before and 3 months after taking Synatura
  The BSS measured cough, sputum, rales/ rhonchi, chest pain during coughing, and dyspnoea. Each of these features of acute bronchitis was scored by a welltrained doctor using a 5point Likert rating scale ranging from 0 to 4 (0 = absent, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe)
  The overall BSS will be graded as mild (0-7), moderate (8-14), and severe (15,20).

CONTACTS AND LOCATIONS:
Overall Officials: Chinkook Rhee, MD, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's hospital, Soeul, South Korea

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2014-11-25): https://cdn.clinicaltrials.gov/large-docs/82/NCT03623282/Prot_000.pdf